CLINICAL TRIAL: NCT00264693
Title: Pharmacokinetics of Dalteparin in Patients With Impaired Renal Function
Status: Completed | Type: Observational
Sponsor: Luzerner Kantonsspital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: W.A. Wuillemin, MD PhD, Head, Division of Hematology and Hematology Central Laboratory, Kantonsspital Luzern, Luzern, Switzerland
Other Study IDs: LMWHplus 3; Ethikkommission Luzern 542; KSL 2006-1H
Record Dates: First submitted 2005-12-11; First posted 2005-12-13 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2009-08

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (8):
- P - A: Prophylactic Dosage, GFR >= 60 mL/min/1.73m^2
- P - B: Prophylactic Dosage, GFR 30-59 mL/min/1.73m^2
- P - C: Prophylactic Dosage, GFR < 30 mL/min/1.73m^2
- P - CAPD: Prophylactic Dosage, CAPD
- T - A: Therapeutic Dosage, GFR >= 60 mL/min/1.73m^2
- T - B: Therapeutic Dosage, GFR 30-59 mL/min/1.73m^2
- T - C: Therapeutic Dosage, GFR < 30 mL/min/1.73m^2
- T - CAPD: Therapeutic Dosage, CAPD

SUMMARY:
Low molecular weight heparins (LMWH) have been shown to be at least as efficient and safe as unfractioned heparin (UFH) in prophylaxis and treatment of venous thromboembolic events and in therapy of acute cardiovascular diseases. LMWH are widely used as safe replacement of oral anticoagulation with vitamin K antagonists (VKA).

Due to their pharmacokinetic characteristics, LMWH tend to accumulate in patients with impaired renal function. Official guidelines recommend therefore to use LMWH controlled by Anti-Xa levels or to use UFH instead of LMWH to provide full therapeutic anticoagulation therapy in patients with severe renal insufficiency.

Although dosage recommendations have been proposed for enoxaparin in patients with renal impairment based on several studies, these data cannot be applied to other LMWH directly due to different pharmacokinetic properties of each drug.

The present study aims to clarify the pharmacokinetics of dalteparin in patients with renal insufficiency, especially addressing the question of accumulation after multiple doses and including patients with severe renal insufficiency and derive a safe and suitable concept for using dalteparin in patients with impaired renal function.

ELIGIBILITY:
Inclusion Criteria:

* Patient starting with dalteparin for prophylaxis OR therapy by order of the treating physician (after having evaluated clinical indication and contraindications).
* Renal function normal OR impaired with or without dialysis therapy according to open study groups
* Age >= 18 years
* Written informed consent

Exclusion Criteria:

* Pregnancy / Lactation
* Dalteparin or other LMWH already in use for > 1 day, unless just in use during hemodialysis
* Anti-Xa level before first application of dalteparin > 0.3 U / ml
* Participation in another study
* Anuria OR glomerular filtration rate < 10 ml/min without dialysis
* Patient on intensive care unit (ICU)
* Cardiovascular unstable patient or probable need for a quick stop of anticoagulation (e.g. emergency surgery)
* Patient with a disease whose estimated life expectancy is < 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of a medical and surcigal department with all levels of renal function who needs Dalteparin for prophylaxis or therapy.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2006-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pirmin Schmid, MD, Principal Investigator — Luzerner Kantonsspital, Hematology; Andreas G Fischer, MD, Study Director — Luzerner Kantonsspital, Nephrology; Walter A Wuillemin, MD, PhD, Study Chair — Luzerner Kantonsspital, Hematology
Locations (1):
- Kantonsspital Luzern, Lucerne, Canton of Lucerne, Switzerland

REFERENCES:
- [Background] Schmid P, Fischer AG, Wuillemin WA. Low-molecular-weight heparin in patients with renal insufficiency. Swiss Med Wkly. 2009 Aug 8;139(31-32):438-52. doi: 10.4414/smw.2009.11284. PMID 19685350
- [Result] Schmid P, Brodmann D, Fischer AG, Wuillemin WA. Study of bioaccumulation of dalteparin at a prophylactic dose in patients with various degrees of impaired renal function. J Thromb Haemost. 2009 Apr;7(4):552-8. doi: 10.1111/j.1538-7836.2009.03292.x. Epub 2009 Jan 19. PMID 19175499
- [Result] Schmid P, Brodmann D, Odermatt Y, Fischer AG, Wuillemin WA. Study of bioaccumulation of dalteparin at a therapeutic dose in patients with renal insufficiency. J Thromb Haemost. 2009 Oct;7(10):1629-32. doi: 10.1111/j.1538-7836.2009.03556.x. Epub 2009 Jul 17. PMID 19624460
- [Result] Schmid P, Brodmann D, Fischer AG, Wuillemin WA. Prospective observational cohort study of bioaccumulation of dalteparin at a prophylactic dose in patients with peritoneal dialysis. J Thromb Haemost. 2010 Apr;8(4):850-2. doi: 10.1111/j.1538-7836.2010.03749.x. Epub 2010 Jan 17. No abstract available. PMID 20088934
- See also: Luzerner Kantonsspital, Hematology — http://www.ksl.ch/standorte/luzern/kliniken/medizin/haematologie.html
- See also: Luzerner Kantonsspital, Nephrology — http://www.ksl.ch/standorte/luzern/kliniken/medizin/nephrologie.html
- See also: Pirmin Schmid — http://www.pirmin-schmid.ch